CLINICAL TRIAL: NCT02437331
Title: National Taipei University of Nursing and Health Science
Brief Title: Experience in Being With Advanced Heart Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201503067RIND
Record Dates: First submitted 2015-04-22; First posted 2015-05-07 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: Advanced heart failure; diseased experience
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- advanced heart failure: the patients was diagnostic on Chronic heart failure with NYHA class 3 and 4, AHA stage D, or LVEF<40%.

SUMMARY:
The purpose of this study is to explore the experience in being with advanced Heart failure patients.

DETAILED DESCRIPTION:
The aim is to explore the experience of advanced Heart failure patients during the disease trajectory in Taiwan.

ELIGIBILITY:
Inclusion criteria:

* the patients' conscious must be clear,
* vital sign is stable,
* and can communicate in Mandarin Chinese or Taiwanese.

exclusion criteria:

* consciousness is unclear
* and can't have effective communication to interviewer.
* the patient reject to join this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study population is diagnosis of advanced heart failure with NYHA class 3 to 4.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
A qualitative research to decribe the experience with advanced Heart failure patients | participants will be followed for the duration of hospital stay, an expected average of 6 weeks.
  describe patterns of diseases traits

CONTACTS AND LOCATIONS:
Overall Officials: keidei kao, master, Principal Investigator — study
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
because the data is still discussing with professional expert. and we think the data is not reach saturation yet.